CLINICAL TRIAL: NCT06807099
Title: Prospective, Multicenter, Observational Study to Evaluate the Merit WRAPSODY® Cell Impermeable Endoprosthesis for Treatment of Stenosis or Occlusion Within the Dialysis Outflow Circuit (WRAP North America)
Brief Title: WRAP North America
Status: Recruiting | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CVO-P4-25-01
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Venous Stenosis; Venous Occlusion
Keywords: Arteriovenous Fistula (AVF); Arteriovenous Graft (AVG); AV fistula; AV graft
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Merit WRAPSODY® Cell Impermeable Endoprosthesis (WRAPSODY CIE) — Target Lesion treated with WRAPSODY CIE

SUMMARY:
The goal of this observational study is to investigate the safety and efficacy of the WRAPSODY CIE in a real-world North American population. Participants treated with the WRAPSODY CIE device in accordance with the device instructions for use will be followed in accordance with standard of care up to 3-years post-procedure.

DETAILED DESCRIPTION:
Prospective, multicenter, observational study to evaluate the Merit WRAPSODY® Cell Impermeable Endoprosthesis for treatment of stenosis or occlusion within the dialysis outflow circuit (WRAP North America)

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent for study participation.
2. Subject is male or female, with an age ≥ 18 years at date of enrollment.
3. Subject is willing to comply with site standard of care procedures and follow-up visit schedules over 36 months.
4. Subject is undergoing chronic hemodialysis with the hemodialysis access the intervention will be performed upon.
5. The dialysis access is considered mature and has been used to deliver hemodialysis treatments for at least one session.
6. Subject has stenosis or occlusion within the dialysis outflow circuit and is treated with WRAPSODY CIE in accordance with device instructions for use.

Exclusion Criteria:

1. Subject has a planned surgical revision of access site.
2. Subject has a known or suspected infection of the hemodialysis access site, systemic infection and/or septicemia.
3. Subject has an uncorrectable coagulation disorder.
4. Known hypersensitivity to nickel or titanium.
5. Subject's hemodialysis access is anticipated to be abandoned within 6 months.
6. Subject is scheduled for kidney transplant or peritoneal dialysis within the next 6 months post-procedure.
7. Full expansion of a PTA balloon cannot be achieved during predilatation.
8. Device would be placed in the Superior Vena Cava
9. Any inflow or outflow lesion that could jeopardize patency access long-term beyond the target treatment area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with stenosis or occlusion within the dialysis outflow circuit who meet the inclusion and exclusion criteria are intended to participate in this study. The eligibility criteria are kept to a minimum to better represent the subject profile treated in actual clinical practice without selecting sub-groups of particular low/high risk or excluding certain diseases or anatomies.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with Target Lesion Primary Patency (TLPP) (Primary Effectiveness Endpoint) | 6 months
  The proportion of subjects with Target Lesion Primary Patency (TLPP) at 6 months.
  Target Lesion Primary Patency (TLPP) defined as freedom from clinically-driven target lesion revascularization (CD-TLR) or target lesion thrombosis measured through 6 months post-procedure, which is the time interval of uninterrupted patency after study procedure to the next intervention performed on the target lesion or uncorrectable target lesion occlusion.
Proportion of subjects without any localized or systemic safety events (Primary Safety Endpoint) | 30 days
  Proportions of subjects without any localized or systematic safety events through 30 days post-procedure that affect the access or venous outflow circuit and resulted in reintervention, hospitalization, or death (not including CD-TLR or target lesion thrombosis)

SECONDARY OUTCOMES:
Proportion of subjects with Target Lesion Primary Patency | 12, 24 and 36 months
  Proportion of subjects with Target Lesion Primary Patency at months 12, 24 and 36.
Proportion of subjects with Assisted Target Lesion Primary Patency (aTLPP) | 6, 12, 24 and 36 months
  Proportion of subjects with Assisted Target Lesion Primary Patency (aTLPP)
Proportion of subjects with Access Circuit Primary Patency (ACPP) | 6, 12, 24 and 36 months
  Proportion of subjects with Access Circuit Primary Patency (ACPP)
Rates of procedure- and device-related adverse events | Index procedure, 30 days, 6, 12, 24 and 36 months
  Number of subjects with procedure- and device-related adverse events

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Medical University of South Carolina, Orangeburg, South Carolina
  - Bluff City Vascular, Memphis, Tennessee
  - Texas Research Institute, Fort Worth, Texas
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No